CLINICAL TRIAL: NCT04373486
Title: Incidence of Acute Pulmonary Embolism in Covid-19 Patients on CT Angiography and Relationship to D-dimer Levels
Acronym: COVID-APE
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7840
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-04

CONDITIONS: Covid-19 With Positive RT-PCR
Keywords: Covid-19; Pulmonary Embolism; CT angiography
MeSH Terms: conditions — COVID-19; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reports of acute pulmonary embolism (APE) associated with COVID-19 have emerged in the literature. For example, Chen et al. described 25 pulmonary CT angiograms examinations from 1008 COVID-19 patients; 10 were positive for pulmonary embolism mostly as segmental or sub-segmental APE. Case reports of APE in Covid-19 patients have been published. Cui et al. found an incidence of deep venous thrombosis in intensive care unit (ICU) patients with severe Covid-19 pneumonia near to 25% (20/81), however without any correlation with potential APE.

Despite these initial reports, it is not clear whether APE is more frequent in Covid-19 patients or if the association is just random. In favor of the former, D-dimer levels have been reported as elevated in patients with Covid-19 by two studies, and it has been suggested an independent association between the severity of the disease and the level of D-dimer. Finally, Tang et al. showed that anticoagulant therapy is associated with a decreased mortality at Day-28 in severe Covid-19 patients, in favor of a possible associated coagulopathy. The purpose of this study is to describe the rate of pulmonary embolus in patients classified as COVID-19 infection and who underwent chest CT angiography.

The purpose of this study is to describe the rate of pulmonary embolus in patients classified as COVID-19 infection and who underwent chest CT angiography.

ELIGIBILITY:
Inclusion Criteria:

* Positive SARS-Cov-2 RT-PCR
* Chest CT angiography available
* Patient is aged 18yo or above

Exclusion Criteria:

* Expressed opposition to participate
* Adults under guardianship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with positive SARS-Cov-2 RT-PCR
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of positivity for Acute Pulmonary Embolism | March 1, 2020 - March 31, 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Radiologie B - NHC, Strasbourg, France